CLINICAL TRIAL: NCT05201560
Title: Efficacy and Safety of Butorphanol Tartrate Injection for the Patients With Mechanical Ventilation:a Randomized and Controlled Trial
Brief Title: Efficacy and Safety of Butorphanol Tartrate Injection for the Patients With Mechanical Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SICU-20211026
Record Dates: First submitted 2021-10-29; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Analgesia; Hospital-acquired Infections
MeSH Terms: conditions — Agnosia | interventions — Butorphanol; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butorphanol tartrate (Experimental): Butorphanol tartrate on the patients with mechanical ventilation
  Interventions: Drug: Butorphanol Tartrate Injection
- fentanyl (Active Comparator): fentanyl on the patients with mechanical ventilation
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Butorphanol Tartrate Injection — Patients of this group will receive Butorphanol Tartrate Injection
  Other Names: the drug of butorphanol tartrate
  Arms: Butorphanol tartrate
Drug: Fentanyl — Patients of this group will receive Fentanyl
  Other Names: the drug of fentanyl
  Arms: fentanyl

SUMMARY:
To compare the incidence of hospital-acquired infections between butorphanol and fentanyl.

DETAILED DESCRIPTION:
Butorphanol can improve inflammation and promote the recovery of pro-inflammatory/anti-inflammatory cytokine balance.However, there is still a lack of relevant clinical studies on butorphanol and fentanyl for the incidence of hospital-acquired infections in ICU mechanically ventilated patients.The objective of this study was to evaluate the analgesic efficacy,safety and the incidence of nosocomial infection of butorphanol in mechanical ventilation patients between butorphanol and fentanyl.

ELIGIBILITY:
Inclusion Criteria:

* need mechanical ventilation for more than 48 hours
* more than 18 years old
* without hospital-acquired infection before admission to ICU
* volunteer to participate in this study

Exclusion Criteria:

* allergic or contraindicated to the drug
* severe cardiac insufficiency, conduction block and bradycardia
* recent use of analgesic, sedative and antidepressant drugs
* psychiatric or neurological diseases or neurosurgery-related diseases
* history of steroid cortisol and immunosuppressants
* severe liver dysfunction or renal dysfunction
* pregnancy
* refuse to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of hospital-acquired infections | one month
  Incidence of hospital-acquired infections

SECONDARY OUTCOMES:
duration on ventilators | one month
  patients enrolled will be followed for the duration of mechanical ventilation
ICU stay | one month
  patients enrolled will be followed for length of ICU stay
Hospital stay | one month
  patients enrolled will be followed for length of Hospital stay
all cause mortality | one month
  all cause mortality
Blood routine examination is assessed by the white blood cell count | on the 1st, 3rd，7th day after enrollment
Blood routine examination is assessed by neutrophil count. | on the 1st, 3rd，7th day after enrollment
Cytokines | on the 1st, 3rd，7th day after enrollment
  Cytokines are assessed by the interleukin-1,interleukin-6 and interleukin-10
adverse events | one month
  Nausea, vomiting, dry mouth, bradycardia, hypotension, respiratory depression and other adverse events

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fridkin SK, Welbel SF, Weinstein RA. Magnitude and prevention of nosocomial infections in the intensive care unit. Infect Dis Clin North Am. 1997 Jun;11(2):479-96. doi: 10.1016/s0891-5520(05)70366-4. PMID 9187957
- [Result] Vincent JL, Rello J, Marshall J, Silva E, Anzueto A, Martin CD, Moreno R, Lipman J, Gomersall C, Sakr Y, Reinhart K; EPIC II Group of Investigators. International study of the prevalence and outcomes of infection in intensive care units. JAMA. 2009 Dec 2;302(21):2323-9. doi: 10.1001/jama.2009.1754. PMID 19952319
- [Result] Meissner W, Dohrn B, Reinhart K. Enteral naloxone reduces gastric tube reflux and frequency of pneumonia in critical care patients during opioid analgesia. Crit Care Med. 2003 Mar;31(3):776-80. doi: 10.1097/01.CCM.0000053652.80849.9F. PMID 12626983
- [Result] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Result] Giamberardino HI, Cesario EP, Carmes ER, Mulinari RA. Risk factors for nosocomial infection in trauma patients. Braz J Infect Dis. 2007 Apr;11(2):285-9. doi: 10.1590/s1413-86702007000200024. PMID 17625779
- [Result] Baviskar AS, Khatib KI, Rajpal D, Dongare HC. Nosocomial infections in surgical intensive care unit: A retrospective single-center study. Int J Crit Illn Inj Sci. 2019 Jan-Mar;9(1):16-20. doi: 10.4103/IJCIIS.IJCIIS_57_18. PMID 30989063
- [Result] Aguilar-Nascimento JE, Marra JG, Slhessarenko N, Fontes CJ. Efficacy of National Nosocomial Infection Surveillance score, acute-phase proteins, and interleukin-6 for predicting postoperative infections following major gastrointestinal surgery. Sao Paulo Med J. 2007 Jan 4;125(1):34-41. doi: 10.1590/s1516-31802007000100007. PMID 17505683